CLINICAL TRIAL: NCT06509165
Title: Comparison of Clinical and Aesthetic Results of Different Techniques in the Treatment of Gingival Recession
Brief Title: Comparison of Different Techniques in the Treatment of Gingival Recession
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Kevser Yildirim, Research Assistant, Necmettin Erbakan University
Other Study IDs: TreatmentofGingivalRecession
Record Dates: First submitted 2024-07-08; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Gingival Recession
Keywords: connective tissue graft; modified coronally advanced flap; tunel technique
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modified coronally advanced flap technique: Patients using a modified coronally placed flap technique to cover gingival recession
  Interventions: Procedure: Modified coronally advanced flap technique
- Tunnel technique: Patients using the tunnel technique to cover gingival recession
  Interventions: Procedure: Tunnel technique

INTERVENTIONS:
Procedure: Modified coronally advanced flap technique — Subepithelial connective tissue graft was applied to the relevant areas with a modified coronally placed flap technique to cover the gingival recession.
  Groups: Modified coronally advanced flap technique
Procedure: Tunnel technique — Subepithelial connective tissue graft was applied to the relevant areas with the tunnel technique to cover the gingival recession.
  Groups: Tunnel technique

SUMMARY:
The aim of this study is to compare the clinical and aesthetic results of different techniques in the treatment of gingival recession.

The main questions it aims to answer are:

* Does the surgical technique preferred by the physician affect the closure rate of gingival recession in the 3rd month?
* Does the surgical technique preferred by the physician affect the closure rate of gingival recession in the 6th month? Participants were informed about the study. Following routine periodontal treatment, surgical operations were performed on the areas with receding gums using different techniques for the patients included in the study.

DETAILED DESCRIPTION:
After the routine clinical and radiological periodontal evaluation of every patient applying to the periodontology department, phase-I periodontal treatment is first applied to every patient diagnosed with periodontal disease. Patients are then given the necessary information to ensure plaque control. Gingival recessions that make mechanical cleaning of the patient difficult and the dentine sensitivity reported by the patient due to these recessions make plaque control difficult for the patient. It is routinely applied to patients who are found to have gingival recessions that cause these problems. These applications vary depending on the withdrawal type.

In patients with gingival recession who apply to the periodontology department, gingival recession closure operations performed with subepithelial connective tissue graft, laterally placed flap, coronally placed flap, modified coronally placed flap, tunnel technique, vestibular incision and subperiosteal tunnel access technique are preferred. The change and recovery status of the patients after the treatments are evaluated and followed up with routine photographs.

Photographs of the procedures and the wound area during and after the operations are taken and stored in the clinic photo archive.

Objective success after root closure procedures is monitored with clinical records and measurements at regular intervals. Success after root closure is evaluated in two categories: clinical and aesthetic success. Clinical success; The reduction in withdrawal depth is determined by measuring clinical binding gain. To determine these, clinical measurements of the patients at the beginning, 1st month, 3rd month, 6th month and 12th month are recorded and photographs are taken. At the same time, since there are other factors that affect both aesthetic and clinical success, the type of recession, aesthetic complaints, sensitivity and brushing effectiveness are recorded before and after treatment. For this reason, the amount of recession, keratinized tissue (mm), clinical attachment level, plaque index, pocket depth, papilla width and height values are recorded and compared in the initial and follow-up examinations of the patients.

Individual choice:

For this study, patients who receive gingival recession treatment at the Periodontology clinic and those who agree to take routine photographs before and after treatment and who sign the consent form if they meet the inclusion criteria for the study will be included. in the study. Our study is a retrospective study. Clinical and photographic records of patients who had previous gingival recession surgery by a clinician at the periodontology clinic will be used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be volunteers between the ages of 18-65,
* Absence of any systemic disease such as impaired glucose tolerance, diabetes mellitus or endocrine disease, nephrotic syndrome, chronic renal disease and cardiovascular disease, Not having used antibiotics in the last 6 months for any reason,
* Not using cigarettes and alcohol,
* Presence of at least 20 teeth in the mouth,
* Not during pregnancy or breastfeeding,
* Not receiving any regulatory drug treatment,
* Patients who applied to the periodontology clinic with various periodontal problems and underwent gingival recession closure surgery using subepithelial connective tissue graft along with modified coronally placed flap and tunnel technique due to the indication of gingival recession.

Exclusion Criteria:

* Being outside the inclusion criteria and not agreeing to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Systemically healthy adults between the ages of 18-65 who applied to the department of periodontology at Necmettin Erbakan University Faculty of Dentistry.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Gingival recession closure amount | 6 months
  How much gingival recession has closed after the operation will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: FATMA UÇAN YARKAÇ, Assoc. Dr., Study Chair — Necmettin Erbakan University Faculty of Dentistry, Department of Periodontology; DİLEK ÖZKAN ŞEN, Asst Prof., Study Director — Necmettin Erbakan University Faculty of Dentistry, Department of Periodontology; ZEYNEP TAŞTAN EROĞLU, Asst Prof., Study Chair — Necmettin Erbakan University Faculty of Dentistry, Department of Periodontology; OSMAN BABAYİĞİT, Asst Prof., Study Chair — Necmettin Erbakan University Faculty of Dentistry, Department of Periodontology; KEVSER YILDIRIM, RESEARCH ASSISTANT, Principal Investigator — Necmettin Erbakan University Faculty of Dentistry, Department of Periodontology
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

REFERENCES:
- [Derived] Yarkac FU, Sen DO, Yildirim K, Eroglu ZT, Babayigit O. Comparison of Clinical and Esthetic Results of Different Techniques in the Treatment of Multiple Gingival Recessions. J Esthet Restor Dent. 2025 Nov;37(11):2358-2367. doi: 10.1111/jerd.70018. Epub 2025 Aug 3. PMID 40755090